CLINICAL TRIAL: NCT05552378
Title: A Single Arm Stuidy to Confirm Safety and Efficacy of Multi-Gyn FloraFem Study for Treatment of Vulvo Vaginal Candidiasis Symptoms
Brief Title: Multi-Gyn FloraFem Study for Treatment of Vulvo Vaginal Candidiasis Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karo Pharma AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22E2054
Record Dates: First submitted 2022-09-20; First posted 2022-09-23 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2022-09

CONDITIONS: Vulvovaginal Candidiasis
MeSH Terms: conditions — Candidiasis, Vulvovaginal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Other)
  Interventions: Device: Multi-Gyn FloraFem

INTERVENTIONS:
Device: Multi-Gyn FloraFem — Vaginal gel packed in 5 single use plastic tubes.

SUMMARY:
Women diagnosed with Vulvovaginal Candidiasis by the health care professional will be enrolled in the study. All participants should fulfil inclusion and exclusion criteria.

The study product will be used for 5 days, once a day. The doctor will evaluate the patients before and at the end of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with Vulvovaginal Candidiasis confirmed by:itching, and/or burning, irritation, edema, redness, crumbly white discharge
* Aged >18 years
* Signed written informed consent form
* Willing to comply to the follow-up schedule
* Subject affiliated to a health social security system.
* Female of childbearing potential should use a contraceptive regimen recognized as effective since at least 12 weeks before screening visit, during all the study and at least 1 month after the study end.

Exclusion Criteria:

* Current clinically manifest of sexually transmitted gynecologically infection, genital tract infection, bacterial vaginosis or aerobic vaginitis (incl. clinical obvious gonorrhoea, chlamydia trachomatis or mycoplasma genitalium infection with cervicitis, urethritis, salpingitis)
* Current genital malignancies
* Chemotherapy for any reason in last 6 months
* Radiotherapy in the genitourinary system in the last 12 months
* Pregnancy or currently attempting to conceive
* Lactation
* Use of other treatment for vaginal conditions during the course of the clinical investigation
* Known allergies to ingredients of the product
* Concomitant medication for treatment of vaginal infections, or other use of intravaginal medication during the course of the clinical investigation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-04-05 (Actual)

PRIMARY OUTCOMES:
To determine the efficacy of Multi-Gyn FloraFem in relieving itch during vaginal candidiasis (based on 0-10 point scale score improvement > 1 related to vulvovaginal candidiasis at Visit 2. | 1 week
  Women should have at least itch related to vaginal candidiasis.

CONTACTS AND LOCATIONS:
Locations (1):
- General Medical Centre, Gdansk, Poland

IPD SHARING:
Plan to Share IPD: No